CLINICAL TRIAL: NCT02267291
Title: Impact of Non-invasive Positive Pressure Ventilation on Cardiac Function and Echocardiographic Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 104/14
Record Dates: First submitted 2014-09-11; First posted 2014-10-17 (Estimated); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Heart Function Tests; Hemodynamics; Noninvasive Ventilation; Circulatory and Respiratory Physiological Phenomena
Keywords: Cardiac Catheterization; Echocardiography; Noninvasive Ventilation; Positive-Pressure Respiration; Ventricular Function

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All patients (Experimental): Ventilatory support to alter intrathoracic pressure
  Interventions: Other: Non-invasive positive pressure ventilation

INTERVENTIONS:
Other: Non-invasive positive pressure ventilation — Ventilatory support to alter intrathoracic pressure

SUMMARY:
Cardiologists and intensive care specialists are confronted daily with mechanically ventilated patients exhibiting cardiac failure. It is of paramount importance to understand the effect of mechanical ventilation on cardiac function and to interpret echocardiographic findings correctly in order to provide the patient with the best possible treatment to support cardiac and circulatory function. Currently physicians interpret echocardiographic findings based on studies that were performed in spontaneously breathing patients. With this study, the investigators intend to contribute to the understanding of cardiac physiology in patients needing ventilatory support, especially they aim to provide the physiological basis for the interpretation of echocardiographic findings in order to improve medical support (e.g. fluid resuscitation, vasoactive drugs, ventilation strategy) of ventilated patients with impaired cardiovascular function.

DETAILED DESCRIPTION:
Background

Mechanical ventilation (MV) is commonly used in intensive care units (ICU) to improve gas exchange and to reduce breathing effort. The need for MV is the single most prominent reason for admission to an intensive care unit, either for acute cardiac or respiratory failure, postoperative ventilation or other reasons. Its usefulness is not limited to critically ill patients but has also gained recognition in treating sleep-related breathing disorders. Soon after the introduction of MV to clinical practice its adverse hemodynamic effects were noted and have been studied ever since. It is now well accepted that MV, by applying external positive pressure in order to achieve tidal breathing, affects lung volume and intrathoracic pressure which in turn influence cardiac loading and function.

Echocardiography is increasingly used in intensive care to evaluate hemodynamics and especially Doppler assessments of mitral inflow and annular tissue velocity to describe left ventricular (LV) diastolic function. There is a growing body of evidence stating that diastolic dysfunction is a key factor for weaning failure from MV, a clinical issue affecting up to one third of patients. Worsened diastolic LV filling under MV may decisively lower cardiac performance and cause hemodynamic instability especially in case of pre-existing diastolic dysfunction in patients with arterial hypertension, a disease with a high prevalence of 30-45% in the general population. So far, despite the extensive use of echocardiography in ventilated patients, the causative pathophysiological mechanisms underlying ventilation-induced changes of echocardiographic parameters used to determine diastolic LV function have never been thoroughly evaluated. Assessing diastolic function during MV is complex since Doppler derived surrogate parameters all depend on cardiac loading conditions and loading itself is inevitably coupled to MV. The question therefore arises whether echocardiography allows for detection of deteriorating LV diastolic function in terms of impaired intrinsic ventricular relaxation or LV stiffness or whether it primarily mirrors MV-induced loading alterations. It is important to differentiate if echocardiographic signs of diastolic dysfunction in the patient under MV are caused by changes in loading or a LV filling restraint since in case of hemodynamic instability the two scenarios would ask for different therapeutic measures. In case of a loading problem, pre- and afterload can be targeted using drugs or fluid resuscitation. If a MV-induced filling restraint is the predominant problem one may consider special ventilatory modes or even deep sedation and the use of muscle relaxants to minimize Pit.

The basic concepts of heart-lung interactions under positive pressure ventilation make it conceivable that extrinsic pressure applied to the thorax and therefore, as explained later in more detail, to the heart may mimic diastolic dysfunction even in a totally healthy heart if assessed by echocardiography. Echocardiographic parameters to assess diastolic function have been evaluated against the gold standard - invasive LV pressure and volume measurements - in spontaneously breathing patients. Such an evaluation is lacking for the patient with ventilatory support and therefore the value of echocardiography for assessment of diastolic function under MV needs further clarification. The investigators intend to comparatively study cardiac and particularly left ventricular diastolic function in ventilated patients using both invasive and ultrasound methods.

Objective

The presented study will elucidate the influence of positive pressure ventilation on cardiac function in humans. Furthermore, the investigators aim to describe the changes of echocardiographic parameters under different levels of positive pressure ventilation and link these changes to the underlying pathophysiological alterations in hemodynamics induced by positive pressure ventilation.

Methods

Prospective single-centre study at the University Hospital Berne. 30 patients scheduled for an elective coronary angiogram will be included. During spontaneous breathing and two different levels of non-invasive PPV transthoracic echocardiography is performed while recording LV-pressure-volume loops using an impedance catheter. Simultaneously the pulmonary artery occlusion pressure, the right atrial pressure and the intrathoracic pressure are recorded using a pulmonary artery catheter and an oesophageal balloon respectively.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 to ≤ 75 years
* Indication for a coronary angiogram
* Written informed consent obtained
* Adequate echocardiographic imaging quality
* • Patient tolerates a face mask for non-invasive ventilation

Exclusion Criteria

* Acute coronary syndrome
* Previous myocardial infarction or open heart surgery
* Severe obstructive or restrictive pulmonary disease
* Pulmonary hypertension
* Diastolic dysfunction ≥ grade II
* Valvular heart disease > grade I
* Left ventricular ejection fraction < 50%
* Complete left or right bundle branch block
* Cardiac pacemaker or defibrillator
* Atrial fibrillation or frequent premature beats
* INR > 3.0 or haemoglobin < 90g/l
* Glomerular filtration rate < 45ml/min/1.73m2
* Esophageal disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Left ventricular diastolic function | Under spontaneous breathing and at two levels of positive pressure ventilation, 5 minutes after changing positive end-expiratory pressure
  Assessed by pressure volume loops

SECONDARY OUTCOMES:
Left ventricular contractility | Under spontaneous breathing and at two levels of positive pressure ventilation, 5 minutes after changing positive end-expiratory pressure
  Assessed by pressure volume loops
Cardiac function | Under spontaneous breathing and at two levels of positive pressure ventilation, 5 minutes after changing positive end-expiratory pressure
  Assessed by echocardiography
Invasively measured alterations in hemodynamics | Under spontaneous breathing and at two levels of positive pressure ventilation, 5 minutes after changing positive end-expiratory pressure
  Alterations of invasively measured hemodynamic parameters including cardiac output and pulmonary artery, right ventricular and right atrial pressures

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Blöchlinger, MD, PhD, Principal Investigator — Department of Cardiology, University Hospital Bern
Locations (1):
- Department of Cardiology, Bern University Hospital, Bern, Canton of Bern, Switzerland

REFERENCES:
- [Derived] Berger D, Wigger O, de Marchi S, Grubler MR, Bloch A, Kurmann R, Stalder O, Bachmann KF, Bloechlinger S. The effects of positive end-expiratory pressure on cardiac function: a comparative echocardiography-conductance catheter study. Clin Res Cardiol. 2022 Jun;111(6):705-719. doi: 10.1007/s00392-022-02014-1. Epub 2022 Apr 6. PMID 35381904